CLINICAL TRIAL: NCT00004793
Title: Pilot Study of the Effect of Baclofen and Bromocriptine on Luteinizing Hormone Secretion in Pubertal Children
Status: Completed | Type: Observational
Sponsor: National Center for Research Resources (NCRR) (NIH)
Collaborators: University of Michigan (Other)
Organization: Office of Rare Diseases (ORD) (NIH)
Other Study IDs: 199/11923; UMMC-1354
Record Dates: First submitted 2000-02-24; First posted 2000-02-25 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2001-12

CONDITIONS: Growth Disorders
Keywords: constitutional growth delay; endocrine disorders; rare disease
MeSH Terms: conditions — Growth Disorders; Puberty, Delayed; Endocrine System Diseases; Rare Diseases

SUMMARY:
OBJECTIVES: I. Evaluate the effect of bromocriptine on luteinizing hormone (LH) secretion by suppression of prolactin and stimulation of dopaminergic receptors in early pubertal boys and girls.

II. Evaluate the effect of baclofen on LH secretion by stimulation of gamma-aminobutyric acid receptors in early pubertal boys and girls.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE:

Participants receive bromocriptine or baclofen followed by nocturnal measurements of luteinizing hormone, growth hormone, and sex steroids. Pituitary reserve is evaluated with the administration of gonadotropin-releasing hormone, and in children undergoing assessment of short stature, standard provocative stimuli.

ELIGIBILITY:
* Short stature and/or constitutional growth delay
* No epilepsy or risk of epilepsy

Ages: 0 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 4
Dates: Start 1995-06

CONTACTS AND LOCATIONS:
Overall Officials: Carol M. Foster, Study Chair — University of Michigan